CLINICAL TRIAL: NCT00871611
Title: Prevalence of Anderson - Fabry Disease in Patients With Left Ventricular Hypertrophy
Brief Title: Viennese Prevalence Study of Anderson-Fabry Disease
Acronym: VIEPAF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Mundigler, Medical University of Vienna
Other Study IDs: VIE190109
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Fabry Disease; Left Ventricular Hypertrophy
Keywords: Hereditary; Anderson-Fabry; prevalence; heart; hypertrophy; urine; globotriaosylceramide; isoforms; α - Galactosidase
MeSH Terms: conditions — Fabry Disease; Hypertrophy, Left Ventricular; Hypertrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
The prevalence of Anderson - Fabry disease in patients with left ventricular hypertrophy is unclear. The investigators will examine urine - α - Galactosidase activity and globotriaosylceramide isoforms in these patients.

DETAILED DESCRIPTION:
Anderson - Fabry disease (AFD) is a rare, X - linked hereditary systemic lysosomal storage disorder which usually affects the heart. The reported incidence of AFD is between 1 in 117000 and 1 in 240000 live births. Due to a deficiency of the enzyme α - galactosidase, glycosphingo-lipids, primarily globotriaosylceramide, are stored also in endothelial and myocardial cells, leading to morphologic and functional changes. AFD-cardiomyopathy progresses with age and with the course of the disease, leading to reduced life expectancy. The investigators hypothesize, that AFD could be underdiagnosed in patients with only mild or moderate left ventricular myocardial hypertrophy. Early diagnosis of AFD may be relevant since affected patients might benefit from enzyme replacement therapy at early stage of disease. The investigators will examine 4000 consecutive patients with an echocardiographically measured interventricular septum thickness of ≥ 12mm. Urine samples will be collected and Gb3-isoforms, creatinine and α - Galactosidase activity will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with myocardial septum wall thickness ≥ 12mm

Exclusion Criteria:

* Patients < 18 years
* Patients unable to provide urine sample

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with left ventricular hypertrophy diagnosed by echocardiography
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Anderson - Fabry disease | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Mundigler, MD, Principal Investigator — Medical University of Vienna, Dept. Internal Medicine, Cardiology
Locations (1):
- Department of Internal Medicine II, Div. Cardiology, Vienna General Hospital, Vienna, Austria

REFERENCES:
- [Background] Weidemann F, Breunig F. [Cardiac involvement in Fabry's disease]. Med Klin (Munich). 2008 Mar 15;103(3):161-5. doi: 10.1007/s00063-008-1023-1. German. PMID 18344066
- [Background] Linhart A, Kampmann C, Zamorano JL, Sunder-Plassmann G, Beck M, Mehta A, Elliott PM; European FOS Investigators. Cardiac manifestations of Anderson-Fabry disease: results from the international Fabry outcome survey. Eur Heart J. 2007 May;28(10):1228-35. doi: 10.1093/eurheartj/ehm153. Epub 2007 May 5. PMID 17483538
- [Background] Monserrat L, Gimeno-Blanes JR, Marin F, Hermida-Prieto M, Garcia-Honrubia A, Perez I, Fernandez X, de Nicolas R, de la Morena G, Paya E, Yague J, Egido J. Prevalence of fabry disease in a cohort of 508 unrelated patients with hypertrophic cardiomyopathy. J Am Coll Cardiol. 2007 Dec 18;50(25):2399-403. doi: 10.1016/j.jacc.2007.06.062. PMID 18154965
- [Background] Fauler G, Rechberger GN, Devrnja D, Erwa W, Plecko B, Kotanko P, Breunig F, Paschke E. Rapid determination of urinary globotriaosylceramide isoform profiles by electrospray ionization mass spectrometry using stearoyl-d35-globotriaosylceramide as internal standard. Rapid Commun Mass Spectrom. 2005;19(11):1499-506. doi: 10.1002/rcm.1948. PMID 15880667